CLINICAL TRIAL: NCT06754085
Title: A Phase III, Prospective, Open-Label, Single-Arm, Multi-center Clinical Study to Assess the Diagnostic Performance and Safety of 18F-Florastamin PET/CT Imaging in Patients With Suspected Recurrence of Prostate Cancer
Brief Title: Study of 18F-Florastamin PET/CT Imaging in Patients With Suspected Recurrence of Prostate Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: HTA Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: BJK-ZX-STM-2203-GK
Record Dates: First submitted 2024-12-23; First posted 2024-12-31 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Injections

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 18F-Florastamin Injection (Experimental)
  Interventions: Drug: Florastamin[18F] Injection

INTERVENTIONS:
Drug: Florastamin[18F] Injection — The subjects will be intravenously injected with a single dose of 7±1 mCi (259±37 MBq) of Florastamin[18F] Injection and undergo PET/CT scan at 60-110 min after the injection.

SUMMARY:
In this study, 18F-Florastamin PET/CT will be performed in patients with suspected recurrence of prostate cancer, to assess the diagnostic performance and safety of 18F-Florastamin PET/CT imaging.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects fully understood the content, process, and potential risks of the study and voluntarily signed an informed consent form (ICF).
2. Male ≥ 18 years of age.
3. Histopathologically confirmed prostate adenocarcinoma per original diagnosis, with subsequent definitive therapy.
4. Suspected recurrence or distant metastasis of prostate cancer based on any of the following conditions:

   1. At least 6 weeks after radical prostatectomy (RP): PSA ≥0.2 ng/mL followed by a subsequent confirmatory PSA value ≥0.2 ng/mL.; or
   2. Post-radiation therapy, after radical radiotherapy (or cryoablation therapy): Increase in PSA level that is elevated by ≥ 2 ng/mL above the nadir .
5. Subjects who are willing to undergo biopsy, salvage surgery, or radiation therapy based on the researcher's clinical judgment;
6. ECOG score 0 or 2.
7. Subjects who meet the following conditions in hematology, renal function, and liver function:

   Platelet count>50 * 10^9/L Urea/urea nitrogen and creatinine<1.5 times upper limits of normal AST and ALT<2.5 times upper limits of normal.
8. Expected survival time ≥ 6 months.
9. Subjects and their partners must use effective contraceptive measurements and avoid sperm donation from the date of signing ICF to 3 months after administration.

Exclusion Criteria:

1. Subjects who have participated in other interventional clinical trials before signing ICF and were within the 5 half-lives of the investigational drug, or who are currently participating in other interventional clinical trials or have participated in clinical trials of radioactive drugs before signing ICF and have been discontinued for less than 3 months until the signing date of ICF.
2. Intravenous injection of iodinated contrast medium within 24 hours, or any high-density oral contrast medium (Such as barium sulfate. Oral water contrast is acceptable, such as compound meglumine diatrizoate oral liquid) within 5 days, prior to study drug administration.
3. Subjects administered any high energy (>300 KeV) gamma-emitting radioisotope within five physical half-lives prior to study drug administration.
4. If previously taking ADT, it should have been discontinued at least 16 weeks prior to study drug administration.
5. The investigator determines that there are any medical diseases or other conditions that affect the safety or compliance of the subjects.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 131 (Estimated)
Dates: Start 2024-12-19 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
The Positive Predictive Value of 18F-Florastamin PET/CT in patients with suspected recurrence of prostate cancer on a patient-level. | 9 months

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, China